CLINICAL TRIAL: NCT00767832
Title: Thromboelastography to Assess Hemostatic Changes in Patients Undergoing Elective Cesarean Delivery.
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Alex James Butwick, Stanford University School of Medicine
Other Study IDs: SU-08252008-1287; 11914
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Venous blood

SUMMARY:
The purpose of the study is to assess the coagulation changes that occur in patients undergoing elective Cesarean delivery using thromboelastography (TEG). We will compare coagulation data to assess potential coagulation changes associated with hemoglobin changes before and after surgery, and related to estimated blood loss.

DETAILED DESCRIPTION:
The purpose of the study is to assess the coagulation changes that occur in patients undergoing elective Cesarean delivery using thromboelastography (TEG). TEG is a point-of-care device which measures the viscoelastic properties of clot formation. This device can provide rapid and detailed information about coagulation changes in the perioperative period. We will compare coagulation data collected from the study to assess potential coagulation changes associated with Hemoglobin changes before and after surgery, and related to estimated blood loss.

ELIGIBILITY:
Inclusion Criteria:

* All obstetric patients with singleton pregnancies admitted to the labor and delivery unit at Lucile Packard Hospital who undergo elective Cesarean delivery.
* We will select 100 healthy ASA 1 patients with singleton pregnancies who are scheduled for uncomplicated elective Cesarean delivery, with no anticipated risk of obstetric hemorrhage.

Exclusion Criteria:

* Patients with underlying coagulation disorders.
* Patients with thrombocytopenia.
* Patients with pregnancy-induced hypertension, pre-eclampsia.
* Patients requiring the following medications prior to surgery: NSAIDS, aspirin, anticoagulants.
* Patients requiring non-elective Cesarean delivery.
* Patients with significant obstetric or medical disease.
* No patients <18 years of age will be recruited.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: healthy pregnant patients undergoing elective cesarean delivery with spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss; Coagulation data (Thromboelastography, Laboratory) | pre and post cesarean delivery

SECONDARY OUTCOMES:
Hematologic indices

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Butwick, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Butwick A, Ting V, Ralls LA, Harter S, Riley E. The association between thromboelastographic parameters and total estimated blood loss in patients undergoing elective cesarean delivery. Anesth Analg. 2011 May;112(5):1041-7. doi: 10.1213/ANE.0b013e318210fc64. Epub 2011 Apr 7. PMID 21474664